CLINICAL TRIAL: NCT05661747
Title: Use of Intraoral Device to Treat Snoring, Sleep Apnea, and Other Symptoms of Sleep-Disordered Breathing in Children
Brief Title: Dental Appliance to Treat SDB in Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vivos BioTechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG-01
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Snoring; Apnea, Obstructive; Upper Airway Resistance Syndrome; Sleep-Disordered Breathing
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: The patient will serve as their own control.
Masking Description: No masking is possible, as each child will serve as their own control in using the mouthguard, and their progress will be compared to their measurements prior to beginning the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention Arm will use Vivos Grow/Vivos Way Device (Experimental): This intervention will compare measurements prior to treatment with measurements post-treatment.
  Interventions: Device: Vivos Grow/Vivos Way Device

INTERVENTIONS:
Device: Vivos Grow/Vivos Way Device — Children already using the device will be monitored to determined whether it improves symptoms of SDB

SUMMARY:
The clinical hypothesis of this study is that a currently marketed mouthguard may also be able to reduce the symptoms of sleep-disordered breathing in children.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of an mouthguard (Vivos Grow/Vivos Way) to reduce sleep-disordered breathing (SDB) in children, including:

snoring, mild to moderate obstructive sleep apnea (OSA), and upper airway resistance syndrome (UARS) in children.

The subjects enrolled in this study will be using the Vivos Grow/Vivos Way to correct orthodontic issues and must also present with signs of SDB.

The study will recruit pediatric subjects who have already elected to utilize the study device for their orthodontic treatment; if they meet the inclusion and exclusion criteria they can be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 6 and under the age of 18 years
* Permanent dentition or mixed dentition at time of evaluation
* Diagnosis of sleep-disordered breathing (including snoring, upper airway resistance syndrome, and/or mild to moderate obstructive sleep apnea)
* Have chosen to have orthodontic treatment
* Living in the United States
* Signed Informed Consent Form

Exclusion Criteria:

* Poor oral hygiene
* Uncontrolled diabetes
* Severe obstructive sleep apnea (AHI> 10/hr)
* Enlarged tonsils of a Grade 4 (>75% of space between pillars)
* Diagnosed with a Temporomandibular join condition (TMJ)
* Any severe breathing or respiratory disorder, such as chronic asthma, emphysema, COPD, or a similar condition
* Orthodontic braces in situ

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pediatric Sleep Questionnaire | An initial evaluation before treatment and upon completion of the study (an average of 1 year)
  Validated questionnaire for determining sleep-related breathing disorders, snoring, and behavior in childrne. The change in score on the PSQ will be assessed. It is scored from 0-1 with higher scores indicating increased symptoms of sleep disturbance and sleep-disordered breathing. Each question is tallied and an average of all answers (from 3 different subsections) gives the final score.
Sleep Study | An initial evaluation before treatment and upon completion of the study (an average of 1 year)
  A home sleep study before and after treatment to assess any changes in sleep disturbance.

SECONDARY OUTCOMES:
Sleep Related Breathing Disordered Questionnaire (SRBD) | An initial evaluation before treatment and upon completion of the study (an average of 1 year)
  A validated subsection of the PSQ, the change in SRBD score will be assessed. It is a 22-questions subset of the PSQ, also graded from 0-1 with scores rising as symptoms of SDB increase.
Airway Volume | An initial evaluation before treatment and upon completion of the study (an average of 1 year)
  Measured using a 3D cone beam scan, the change in airway volume will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Musso, DDS, Principal Investigator — Musso Family Dentistry
Locations (4):
- United States (4):
  - Breathing and Sleep Center, Colorado Springs, Colorado
  - Emerald Coast Dental Spa and Sleep Medicine, Panama City Beach, Florida
  - Musso Family Dentistry, Garland, Texas
  - New Teeth Dental Solutions, League City, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kushida CA, Stevens J, Bennett M, Heit T, Klemp D, Raio D, Cozean J, Cozean C. Multicenter clinical trial for the treatment of obstructive sleep apnea with a non-permanent orthodontic intraoral device in children. Eur J Pediatr. 2025 Jun 17;184(7):424. doi: 10.1007/s00431-025-06254-x. PMID 40526156